CLINICAL TRIAL: NCT06718933
Title: A Prospective, Single-arm, Exploratory, Phase Ib/II Study of SHR-A1811 Combined With Pyrotinib and Bevacizumab in Advanced Breast Cancer With Brain Metastasis.
Brief Title: Study of SHR-A1811 Combined With Pyrotinib and Bevacizumab in Advanced Breast Cancer With Brain Metastasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief physician, Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCBM-004
Record Dates: First submitted 2024-11-20; First posted 2024-12-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Metastatic; Breast Cancer Brain Metastases
MeSH Terms: interventions — Bevacizumab; pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHR-A1811+pyrotinib (Experimental): In phase Ib, enrolled subjects will received SHR-A1811 combined with pyrotinib at different doses to confirm RP2D and evaluate the safety and tolerance.
  Interventions: Drug: SHR-A1811; Drug: Pyrotinib
- SHR-A1811+pyrotinib+bevacizumab (Experimental): In phase II, enrolled subjects will received SHR-A1811 combined with pyrotinib and bevacizumab to evaluate the efficacy and safety.
  Interventions: Drug: SHR-A1811; Drug: Bevacizumab; Drug: Pyrotinib

INTERVENTIONS:
Drug: SHR-A1811 — ADC
Drug: Bevacizumab — bevacizumab biosimilar
  Arms: SHR-A1811+pyrotinib+bevacizumab
Drug: Pyrotinib — anti-HER2 inhibitor

SUMMARY:
In phase Ib, our study is aimed to evaluate the safety and tolerance of SHR-A1811 combined with pyrotinib in breast cancer with brain metastasis, and confirm the recommended phase 2 dose combined with preliminary results of efficacy.

In phase II, our study is aimed to evaluate the efficacy and safety of SHR-A1811 combined with pyrotinib and bevacizumab at RP2D in breast cancer with brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old;
* ECOG PS Score: 0~2;
* Patients must have a life expectancy ≥ 3 months;
* Brian metastasis confirmed by MRI, at least one measurable brain lesion based on RANO-BM with no prior radiotherapy;
* Mannitol or hormone therapy is allowed to use for brain metastasis before enrolment, but treatment dosage should be stable for one week and not need to be increased;
* Adequate organ function and marrow function;
* Has recovered from any AEs (≤ grade 1) related to prior anti-tumour treatments before first dose of study therapy, except: a. alopecia; b. hyperpigmentation;
* Willing to join in this study, able to provide written informed consent, good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

* Has leptomeningeal metastasis or cystic metastatic lesions confirmed by MRI or lumbar puncture;
* Existence of third space fluid (e.g. massive ascites, pleural effusion, pericardial effusion) that is not well controlled by effective methods, e.g. drainage;
* Has CNS complications with the need for emergency intervention, or brain metastasis with poorly controlled symptoms by hormone or dehydration therapy, such as uncontrollable intracranial hypertension, mental disorder or epilepsy;
* Prior bevacizumab or EGFR-TKI is allowed, but should meet the following requirements at the same time:

  1. No disease progression during prior bevacizumab or EGFR-TKI;
  2. More than 3 months from the interruption of bevacizumab or EGFR-TKI to disease progression;
* Has received whole brain radiotherapy, chemotherapy, surgery within 2 weeks before first dose of study therapy; has received trastuzumab-based therapy or endocrine therapy within one week before first dose of study therapy; has received palliative radiotherapy for bone metastasis within 2 weeks before first dose of study therapy;
* Has known clinically significant lung disease, that is, moderate-to-severe lung disease which severely affects respiratory function, including but not limited to: idiopathic pulmonary fibrosis, pneumonitis. Prior ≥ grade 3 interstitial lung disease is not allowed to enrolment;
* Has received full-dose anticoagulants or thrombolytics within 10 days before enrolment, or non-steroid anti-inflammatory drugs with platelet inhibition (except low-dose aspirin (≤325mg qd) for preventive use);
* Existence of unhealed wound, active gastric ulcer, and other diseases which may cause haemorrhage risk (e.g., prior major operation within 4 weeks before enrolment, prior arterial or venous thrombotic event within one year before enrolment, prior cerebralvascular accident);
* Has known hereditary haemorrhagic tendency or coagulation disorder;
* Has joined in other clinical drug trials within 2 weeks before enrolment;
* Use of other antitumor systemic treatment during the study at the same time, except bisphosphonates for the treatment of bone metastasis or osteoporosis prevention;
* Other malignancy within prior 5 years unless curatively treated with no evidence of disease for at least recent 3 years, except: curatively treated in situ cancer of the cervix, skin basal cell carcinoma or skin squamous cell carcinoma;
* Cardiac insufficiency, including but not limited to: congestive heart failure, transmural myocardial infarction, angina which needs drug treatments, clinically significant valvulopathy and high-risk arrhythmia, or QTc abnormity with clinical significance in ECG examination during the screening period (corrected QTc >450 msec [male] or QTc >470 msec [female] under the resting state);
* Uncontrolled hypertension (under the resting state: systolic pressure >160mmHg or diastolic pressure >100mmHg);
* Other diseases which may affect study results, including but not limited to: 1) known history of immunodeficiency, including HIV-positive, other acquired or innate immunodeficient disease, or known history of organ transplantation; 2) HBsAg-positive and HBV DNA≥1000 IU/mL, or HCV antibody-positive, or treponema pallidum antibody-positive; 3) hypersensitivity to study therapy or any of its excipients; 4) severe infection requiring antibiotics, antiviral or antifungal treatment;
* Female patients during the gestation or suckling period, of childbearing potential and pregnancy test-positive, or unwilling to use an effective method of contraception during the whole study;
* Inability to swallow, intestinal obstruction or existence of other factors affecting medication and absorption;
* Any other conditions not appropriate for study enrolment in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
RP2D in phase Ib | From the enrolment of the first subject, to the end of Cycle 6 completion or disease progression or dose discontinuation due to AE in the last enrolled subject
  Recommended phase II dose confirmed by maximum tolerated dose (MTD) and tolerance of subjects.
CNS-ORR by investigator in phase II | At baseline, at the time point of every 6 weeks
  CNS-ORR is the percentage of evaluable patients with a confirmed investigator-assessed CNS response of CR (complete response) or PR (partial response) per RANO-BM.

SECONDARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) in phase Ib | At the time point of 21 days from first medication
  Incidence of DLT
MTD in phase Ib | From the enrolment of the first subject, to the end of Cycle 6 completion or disease progression or dose discontinuation due to AE in the last enrolled subject
  MTD is the highest dose that does not cause any adverse effects as follows: a) 1 subject experienced the treatment-related serious adverse effects that could endanger the life, cause permanent disability or death; b) 2 of 3 subjects experienced DLTs; c) 1 of the first 3 subjects experienced DLTs, and 1 of the additional 3 subjects at the same dose level experienced DLTs again.
Incidence and grade of adverse event (AE) and serious adverse event (SAE) in phase Ib | From the time of informed consent provided to 3 months after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. An SAE is defined as any medical event that results in any of the following outcomes: requires inpatient hospitalization or prolongation of existing hospitalization, disability or incapacity, affects ability to work, a life-threatening adverse event or death, a congenital anomaly.
CNS-ORR per RANO-BM in phase Ib | At baseline, at the time point of every 6 weeks
  CNS-ORR is the percentage of evaluable patients with a confirmed CNS response of CR (complete response) or PR (partial response) per RANO-BM.
CNS-ORR per RECIST v1.1 in phase Ib | At baseline, at the time point of every 6 weeks
  CNS-ORR is the percentage of evaluable patients with a confirmed CNS response of CR (complete response) or PR (partial response) per RECIST v1.1.
CNS-DCR in phase Ib | At baseline, at the time point of every 6 weeks
  CNS-DCR is the percentage of evaluable patients with a confirmed CNS response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1.
DoR in phase Ib | up to 2 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
CNS-ORR per RECIST v1.1 in phase II | At baseline, at the time point of every 6 weeks
  CNS-ORR is the percentage of evaluable patients with a confirmed CNS response of CR (complete response) or PR (partial response) per RECIST v1.1.
CNS-DCR in phase II | At baseline, at the time point of every 6 weeks
  CNS-DCR is the percentage of evaluable patients with a confirmed CNS response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1.
DoR in phase II | up to 2 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
PFS in phase II | up to 2 years
  PFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression).
OS in phase II | up to 2 years
  OS is the time from the date of first dose until the date of death by any cause.
Safety in phase II | From the time of informed consent provided to 30 days after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Chief physician, Principal Investigator — Fudan University; Biyun Wang, Chief physician, Principal Investigator — Fudan University
Locations (1):
- Fudan Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No